CLINICAL TRIAL: NCT04584892
Title: Turoctocog Alfa in Haemophilic Italian Patients: Protection and Engagement in Recreational Activities (THIRd). An Observational, Prospective, Multicentre, Cohort Study on Italian Patients With Haemophilia A in Prophylaxis Treatment With Turoctocog Alfa Under Current Clinical Conditions
Brief Title: Turoctocog Alfa in Haemophilic Italian Patients: Protection and Engagement in Recreational Activities
Acronym: THIRd
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7008-4655; U1111-1247-5494 (Other: World Health Organisation (WHO))
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemophilia A: Patients enrolled will have Haemophilia A (any severity), needing turoctocog alpha prophylactic therapy.
  Interventions: Drug: Turoctocog alfa

INTERVENTIONS:
Drug: Turoctocog alfa — Patients will be treated with commercially available NovoEight® (turoctocog alfa) according to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available NovoEight® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
This is a study on Italian patients with haemophilia A in prophylaxis treatment with Turoctocog alfa under routine clinical conditions. The purpose of the study is to investigate the therapeutic scheme in a population of patients treated with Turoctocog alfa and to investigate the participation in recreational activities, the level of physical activity, and quality of life. Participants will get NovoEight® (Turoctocog alfa) as prescribed to them by the study doctor. The study will last for about 12 months. Participants will be requested to fill in the Questionnaires investigating the participation in recreational activities, the level of physical activity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age above or equal to 12 years at the time of signing informed consent.
* Haemophilia A (any severity), needing prophylactic therapy (with the usual recommended doses).
* Decision to treat with turoctocog alfa, made by the treating Physician and the subject/Legally Acceptable Representative (LAR) based on local label before and independently from the decision to include the subject in this study.

Exclusion Criteria:

* Previous participation in this study, defined as previously signed informed consent;
* Presence of other coagulation disorders;
* Presence of any inhibitor;
* Mental problems, poor compliance, linguistic barriers or other conditions which can impede the understanding of the study aims and the participation to it.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled will have Haemophilia A (any severity), needing turoctocog alpha prophylactic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Individual prophylaxis (PPX) regimen with turoctocog alfa: Every second day, or three times a week (3TW), or twice a week (2TW) | Baseline (week 0)
  Count

SECONDARY OUTCOMES:
Individual PPX regimen with turoctocog alfa: every second day, or 3TW, or 2TW | Final visit (12 months)
  Count
Change of PPX regimen: YES/NO | 12 months after treatment initiation
  Count (participants who have changed regimen or not)
Reported reasons for change of PPX regimens | Final visit (12 months)
  Count (reasons according to the predefined list, see below)
  Individual reported reasons for switch will be selected among the following predefined:
  1. to improve articular protection
  2. due to bleedings
  3. due to patients' needs, including: physical inactivity, work, recreational activity, travel, other.
Difference in score of 'Bridging Hemophilia Experiences, Results, and Opportunities' BHERO questionnaire | Final visit (12 months) vs Baseline (week 0)
  Points
  The following sections of the BHERO questionnaire will be used:
  1. Haemophilia Activities List (HAL: measures the impact of haemophilia on self-perceived functional abilities in patients (42 questions in 7 domains). Scores from 1 (worst) to 6 (best). The final score is the sum of all the scores.)
  2. Recreational and sport activities
  3. Brief pain inventory, exploring the presence and intensity of physical pain, and its impact on performance of daily activities.
  4. International Physical Activities questionnaire (IPAQ) score (Score<700 = Inactive Patient, Score 700 to 2519 = Sufficiently active patient, Score ≥ 2520 = Active or very active patient.
Difference in circulating turoctocog alfa levels | Final visit (12 months) vs Baseline (week 0)
  IU/mL
  Before 12 months visit, monitoring will be reported only if measured in clinical practice due to bleedings or other clinical reasons.
Individual Annual Bleeding Rate (ABR) | From baseline to final visit (12 months)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (10):
- Italy (10):
  - Novo Nordisk Investigational Site, Milan, MI
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Castelfranco Veneto
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Cesena
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Vicenza

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com